CLINICAL TRIAL: NCT00950911
Title: An Open Label, Single Arm, Extension Study to Evaluate the Long Term Safety of Denosumab in the Treatment of Bone Metastases in Subjects With Advanced Cancer or Multiple Myeloma
Brief Title: Open Label Extension to SRE Studies in United Kingdom and Czech Republic Only
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20080540
Record Dates: First submitted 2009-07-30; First posted 2009-08-03 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2013-12

CONDITIONS: Bone Metastases in Men With Hormone-Refractory Prostate Cancer; Bone Metastases in Subjects With Advanced Breast Cancer; Bone Metastases in Subjects With Advanced Cancer or Multiple Myeloma
Keywords: Bone metastases; Hormone-refractory prostate cancer; Multiple myeloma; Denosumab; Breast cancer; 20050103; 20050136; 20050244; Advanced cancer; Tumor; Prostate cancer; Zoledronic acid
MeSH Terms: conditions — Multiple Myeloma; Breast Neoplasms; Neoplasms; Prostatic Neoplasms | interventions — Denosumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: amg 162

INTERVENTIONS:
Drug: amg 162 — 120 mg SC injection of denosumab Q4W until the subject has access to commercially available product or for up to 2 years, which ever comes first.

SUMMARY:
The purpose of this study is to describe the safety and tolerability of denosumab administration as measured by adverse events, immunogenicity, and safety laboratory parameters in subjects who previously received either zoledronic acid (Zometa®) or denosumab.

ELIGIBILITY:
Inclusion Criteria:

* Subjects currently enrolled in study 20050103, 20050136, or 20050244
* Subjects must sign the informed consent before any study specific procedures are performed

Exclusion Criteria:

* Developed sensitivity to mammalian cell derived drug products during the 20050103, 20050136, or 20050244 study
* Currently receiving any unapproved investigational product other than denosumab
* Subject is pregnant or breast feeding, or planning to become pregnant within 7 months after the end of treatment
* Subject (male or female) is not willing to use 2 highly effective contraception during treatment and for 7 months (women) or 10 months (men) after the end of treatment
* Male subject with a pregnant partner who is not willing to use a condom during treatment and for additional 10 months after the end of treatment
* Any disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-07; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (12):
- Czechia (5):
  - Research Site, Jindřichův Hradec
  - Research Site, Kroměříž
  - Research Site, Olomouc
  - Research Site, Prague
  - Research Site, Zlín
- United Kingdom (7):
  - Research Site, Chichester
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Northwood
  - Research Site, Peterborough
  - Research Site, York

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recuited in this open-label extension study were those who were enrolled in the 2 parent (phase 3, randomized, double-blind, active-controlled) studies 20050103 (NCT00321620) or 20050136 (NCT00321464) at sites in the Czech Republic and United Kingdom.
Groups:
- Zoledronic Acid 4 mg Q4W / Denosumab 120 mg Q4W: This cohort received Zoledronic Acid 4 mg Q4W in the blinded treatment phase of the parent study 20050103 (NCT00321620) or 20050136 (NCT00321464), and received Denosumab 120 mg Q4W in this open-label extension study.
- Denosumab 120 mg Q4W / Denosumab 120 mg Q4W: This cohort received Denosumab 120 mg Q4W in the blinded treatment phase of the parent study 20050103 (NCT00321620) or 20050136 (NCT00321464), and received Denosumab 120 mg Q4W in this open-label extension study.
Period: Overall Study
Arm/Group | Zoledronic Acid 4 mg Q4W / Denosumab 120 mg Q4W | Denosumab 120 mg Q4W / Denosumab 120 mg Q4W
Started | 17 | 18
Completed | 5 | 3
Not Completed | 12 | 15
Not completed — Adverse Event | 0 | 2
Not completed — Death | 4 | 6
Not completed — Disease progression | 2 | 2
Not completed — Consent withdrawn | 1 | 3
Not completed — Administrative decision | 3 | 1
Not completed — Ineligibility determined | 1 | 0
Not completed — Noncompliance | 1 | 0
Not completed — Poor performance status | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid 4 mg Q4W / Denosumab 120 mg Q4W | Denosumab 120 mg Q4W / Denosumab 120 mg Q4W | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (11.1) | 61.1 (13.0) | 61.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 10 | 12 | 22
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 17 | 17 | 34
  Black or African American | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Survived
Time Frame: 2 years
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid 4 mg Q4W / Denosumab 120 mg Q4W | Denosumab 120 mg Q4W / Denosumab 120 mg Q4W
Number analyzed (Participants) | 17 | 18
Participants | 13 | 12

ADVERSE EVENTS:
Time Frame: 2 years
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Zoledronic Acid 4 mg Q4W / Denosumab 120 mg Q4W | Denosumab 120 mg Q4W / Denosumab 120 mg Q4W
Serious Adverse Events (participants affected / at risk) | 8/17 | 10/18
Other Adverse Events (participants affected / at risk) | 13/17 | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 4 mg Q4W / Denosumab 120 mg Q4W (N=17) | Denosumab 120 mg Q4W / Denosumab 120 mg Q4W (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 4 mg Q4W / Denosumab 120 mg Q4W (N=17) | Denosumab 120 mg Q4W / Denosumab 120 mg Q4W (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 | 6
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0
Cushingoid (Endocrine disorders) | 1 | 1
Eye pain (Eye disorders) | 1 | 0
Eye swelling (Eye disorders) | 1 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Gingivitis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 5
Oral disorder (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 2
Tooth loss (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3
Chest pain (General disorders) | 2 | 0
Face oedema (General disorders) | 1 | 0
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 6
Feeling hot (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 2
Local swelling (General disorders) | 1 | 0
Localised oedema (General disorders) | 1 | 0
Mucosal necrosis (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 0
Pain (General disorders) | 2 | 2
Pyrexia (General disorders) | 1 | 0
Submandibular mass (General disorders) | 0 | 1
Swelling (General disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Immunodeficiency (Immune system disorders) | 1 | 0
Borrelia infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 2
Oral fungal infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 2
Periostitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Coordination abnormal (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 2 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 1 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 2
Paraesthesia (Nervous system disorders) | 2 | 2
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Penile oedema (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity allergic reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Denture wearer (Social circumstances) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.